CLINICAL TRIAL: NCT02250625
Title: A Prospective Collection of Peripheral Blood Specimens to Study Vitamin D in Healthy Individuals
Brief Title: Study Vitamin D in Healthy Individuals
Status: Completed | Type: Observational
Sponsor: Fujirebio Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FDI-88
Record Dates: First submitted 2014-09-24; First posted 2014-09-26 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
To obtain sufficient specimens and correlating clinical data from a well-controlled prospective clinical trial collecting specimens from healthy subjects t on vitamin D assays, and to establish a collection of specimens that will support future assay discovery and validation efforts.

DETAILED DESCRIPTION:
1. Obtain matched serum and plasma specimens collected from a minimum of 50 healthy subjects in two geographic areas. Specimens will be used to determine a reference range for a vitamin D assay, used as an aid in the assessment of vitamin D sufficiency in adults.
2. Obtain serum specimens collected from a minimum of an additional 450 healthy subjects in two geographic areas. Specimens will be used to determine a reference range for a vitamin D assay, used as an aid in the assessment of vitamin D sufficiency in adults.
3. To store any remaining specimens for use in future vitamin D assay development and to evaluate as yet undetermined assays for the development of IVDs, including additional vitamin D assays

ELIGIBILITY:
Inclusion Criteria:

Males and females, age≥ 18 years Able to understand and willing to provide informed consent

Exclusion Criteria:

Males and females, age <18 years Current use of dietary supplements (tablet, liquid gel or liquid form only) containing high concentrations, greater than 2,000 IU per day, of vitamin D.

Has a history of vitamin D deficiency Has a history or current diagnosis of any clinically significant cardiac, respiratory, neurological, immunological, hematological, liver disease, renal disease, gastrointestinal (GI) disorder, including any history of peptic or gastric ulcers or GI bleeding, or any other condition which, in the opinion of the investigator is considered chronic.

Personal history of seizures Personal history of bariatric surgery Personal history of parathyroid and thyroid disease Pregnancy or lactation Is receiving systemic chemotherapy or radiation treatment, has an active malignancy of any type, or has been diagnosed with cancer within 5 years before screening other than basal or squamous cell skin cancers or in-situ cervical cancer.

Family history of parathyroid or calcium regulatory disease Medications known to affect absorption e.g. drugs that inhibit cholesterol absorption Medications known to increase catabolism such as anticonvulsants, glucocorticoids, HAART (AIDS treatment) and anti-rejection medications Unable to provide informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy men and women greater than or equal to 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 482 (Actual)
Dates: Start 2014-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Measure Vitamin D in healthy individuals | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kogelnik, MD,PhD, Principal Investigator — Open Medicine Institute
Locations (1):
- Open Medicine Institute, Mountain View, California, United States